CLINICAL TRIAL: NCT00730899
Title: Observational Association Study of G Protein Polymorphisms With Cardiac Performance in Coronary Artery Disease Patients Undergoing Coronary Artery Bypass Grafting
Brief Title: Association Study of Gene Polymorphisms With Cardiac Performance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Ulrich Frey, University Hospital Essen
Other Study IDs: HOT-001
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Genetic Polymorphism; Coronary Artery Disease; Hemodynamics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether polymorphisms in G protein subunits, namely Galphas and Galphaq, are associated with altered cardiac performance in heart failure patients.

DETAILED DESCRIPTION:
G Protein pathways plays a pivotal role in mediating positive inotropy and cardiac hypertrophy by transducing signals of neurohormones in cardiomyocytes. Single nucleotide polymorphisms (SNPs) in the G protein subunits Galphas and Galphaq have been shown to result in altered protein expression. We now want to examine whether G Protein polymorphisms alter NYHA functional class, and hemodynamic variables in patients with coronary artery disease scheduled for coronary artery bypass grafting .

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of coronary artery disease
* patients scheduled for coronary artery bypass grafting

Exclusion Criteria:

* emergency operation
* combined vitium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease scheduled for coronary artery bypass grafting in the university hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-01 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
genotype dependent change of hemodynamic variables | one day

SECONDARY OUTCOMES:
all cause mortality | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Peters, MD, Study Director — University Hospital, Essen
Locations (1):
- University Hospital, Essen, North Rhine-Westphalia, Germany